CLINICAL TRIAL: NCT07354698
Title: Application of Mitoxantrone Hydrochloride Injection in Transoral Robotic Thyroid Cancer Surgery
Acronym: MHI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: No.08[2024]; No.08[2024] (Other: DapingH)
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Papillary Thyroid Cancer
Keywords: Mitoxantrone Hydrochloride Injection; Transoral Robotic Surgery
MeSH Terms: conditions — Thyroid Cancer, Papillary | interventions — Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mitoxantrone Hydrochloride Injection (Experimental): The experimental group used mitoxantrone hydrochloride injection as a lymphatic tracer to distinguish the parathyroid glands and lymph nodes according to the blue staining during the operation.
  Interventions: Drug: mitoxantrone hydrochloride injection
- the blank control group (No Intervention): the blank control group does not receive any tracers, and the operating surgeon distinguishes the parathyroid glands and lymph nodes with the naked eye with experience, anatomy, etc.

INTERVENTIONS:
Drug: mitoxantrone hydrochloride injection — The experimental group used mitoxantrone hydrochloride injection as a lymphatic tracer to distinguish the parathyroid glands and lymph nodes according to the blue staining during the operation.
  Arms: Mitoxantrone Hydrochloride Injection

SUMMARY:
Dear Patient, You are invited to participate in a clinical study investigating the Application of Mitoxantrone Hydrochloride Injection for Lymphatic Tracing in Transoral Robotic Thyroid Cancer Surgery. This protocol (Protocol No.: [To be filled]) has been reviewed and approved by the Ethics Committee of the Army Center of Specialized Medicine.

I. Background and Objectives 1.1 Disease Burden and Current Treatments 1.1.1 Thyroid Cancer Surgery Thyroid cancer, the most common head and neck malignancy, exhibits rising global incidence. Central compartment lymph nodes are frequent sites of metastasis in papillary thyroid carcinoma (PTC). Transoral endoscopic thyroid surgery offers superior cosmesis versus open surgery. The da Vinci® robotic system enhances visualization and instrument maneuverability, overcoming technical limitations of narrow endoscopic operating channels.

1.1.2 Lymphatic Tracers in Thyroid Surgery

Mitoxantrone Hydrochloride Injection for Lymphatic Tracing is China's only approved tracer for thyroid lymphatic mapping. Its high lymphotropic specificity enables:

Lymph node mapping: Forms nanocrystals that permeate lymphatics, staining nodes blue.

Parathyroid negative imaging: Spares parathyroid glands, aiding their identification and reducing postoperative hypocalcemia.

1.2 Study Objectives

Primary: Compare lymph node dissection efficacy and parathyroid protection between:

Intervention: Transoral robotic thyroid lobectomy/total thyroidectomy + central neck dissection (CND) with lymphatic tracing.

Control: Identical surgery without tracing.

Secondary:

1. Compare postoperative parathyroid function between groups.
2. Evaluate tracer sensitivity for metastatic lymph nodes.

1.3 Participating Site and Sample Size Site: Army Center of Specialized Medicine Sample: 114 treatment-naïve PTC patients scheduled for transoral robotic surgery (Jan-Dec 2024).

Intervention group (n=57): Mitoxantrone Hydrochloride tracing Control group (n=57): No tracer II. Study Procedures Pre-study: Medical history review, preoperative assessments, and documentation of concomitant medications (30 days postsurgery).

Intervention:

Thyroid exposure → Intervention group: Multisite intraglandular tracer injection (0.1 mL/site, depth ≈0.3 cm; total dose thyroid-dependent).

Both groups: Thyroid lobectomy/total thyroidectomy ± unilateral/bilateral CND. Intraoperative recording: Thyroid characteristics, tracer dose/injection sites, lymphadenectomy duration.

Pathology:

Total lymph node yield and blue-staining rate. Intraoperative frozen section + final histopathology for metastatic nodes.

Follow-up (Postoperative Day 7±3):

Physical exam, vital signs, lab tests (CBC, biochemistry, thyroid/parathyroid hormones, electrolytes).

12-lead ECG. Safety monitoring: Adverse events (AEs) tracked until Postoperative Day 14. III. Potential Benefits Improved lymphatic mapping → Reduced parathyroid injury, enhanced lymph node clearance, lower AE rates.

Tracer provided at no cost by the sponsor. Note: Efficacy is not guaranteed. Alternative treatments exist. IV. Risks and Inconveniences Potential AEs: Per product labeling and surgical risks. Procedural burdens: Multiple hospital visits and tests. AE management: Immediate medical intervention provided. Compensation per GCP regulations if injury is trial-related.

V. Costs Tracer: NMPA-approved and insurance-covered. Routine care/medications: Patient/insurance responsibility. AE compensation: Sponsor-covered if causally related (per Chinese GCP). VI. Confidentiality

Medical records accessible only to:

Research team Ethics Committee Regulatory authorities No personally identifiable data will be published. VII. Contact Information Ethics Committee: 68757140 Principal Investigator: Dr. Yan Xu / TEL: 68729250 VIII. Voluntary Participation Right to withdraw anytime without penalty. Investigator may discontinue your participation for safety/administrative reasons.

Exit assessments may be required. IX. Decision Process Discuss with your physician/family. Retain this document.

Participant Signature: ___________________ Date: _________

Investigator Signature: ___________________ Date: _________

DETAILED DESCRIPTION:
1. Incidence of hypoparathyroidism
2. Positive lymph node tracing rate

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old, both male and female;
* Preoperative neck ultrasound and/or puncture pathology suggested thyroid cancer, and postoperative pathology diagnosed thyroid cancer (tumor diameter <4cm);
* There are no obvious contraindications to surgery during routine preoperative examination;
* Meet the indications for thyroid lobe/total resection + unilateral/bilateral central lymph node dissection;
* Subjects voluntarily join this study, sign the informed consent form, have good compliance, and cooperate with follow-up. 4.2 Exclusion Criteria

Exclusion Criteria:

* Those who have a history of severe drug allergy or are allergic to the drugs in this study;
* Those with serious primary diseases such as cardiovascular and cerebrovascular, liver, kidney, and hematological system;
* Combined with parathyroid disease or other calcium and phosphorus metabolism-related diseases;
* Benign thyroid lesions;
* Received mitoxantrone treatment within 4 weeks;
* Enrolled in other clinical studies at the same time;
* Known history of psychotropic drug abuse, alcohol abuse or drug abuse;
* Pregnant or lactating women;
* According to the investigator's judgment, the subject has other factors that may cause him to be forced to terminate the study midway, such as suffering from other serious diseases (including mental illness) requiring combined treatment, serious abnormal laboratory examination values, family or social factors, which may affect the safety of the subject or the collection of trial data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of parathyroid missections | 1week
  Number of parathyroid missections

SECONDARY OUTCOMES:
Number of lymph node dissections in the central region | 2week
  Number of lymph node dissections in the central region

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Chongqicun, China

IPD SHARING:
Plan to Share IPD: No
The study is confidential and the study data is not open to the public

REFERENCES:
- Available data/document: Individual Participant Data Set: Daping H — http://www.dph-fsi.com/ — Mitoxantrone Hydrochloride Injection